CLINICAL TRIAL: NCT05220605
Title: Safety of Nebulised Delivery of BromAc® (Bromelain & Acetylcysteine) in Healthy Volunteers: a Potential Treatment for Severe COVID-19
Brief Title: Nebulised BromAc in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mucpharm Pty Ltd (Industry)
Collaborators: St George Hospital, Australia (Other); Mobius Medical Pty Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MUC-COV-002
Record Dates: First submitted 2022-01-24; First posted 2022-02-02 (Actual); Last update posted 2022-09-15 (Actual); Status verified 2022-09

CONDITIONS: COVID-19 Pneumonia; Bromelains Adverse Reaction; Acetylcysteine Adverse Reaction; Mucus; Plug; COVID-19 Acute Respiratory Distress Syndrome
Keywords: bromelain; BromAc; acetylcysteine; SARS-CoV-2; mucin; mucus plug; COVID-19 pneumonia; ventilator associated pneumonia; secondary bacterial infection
MeSH Terms: conditions — Medullary cystic kidney disease 1; Pneumonia, Ventilator-Associated | interventions — bromelain and acetylcysteine drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Bromac (100ug/20mg) (Experimental): The nurse/investigator will fill the jet nebuliser canister supplied on the ward with the 5ml of BromAc (100micrograms bromelain and 20mg acetylcysteine). The cannister will be collected to the mask and attached to the wall compressed air supply, with flow of between 6-8L per minute. The mask will be placed on the participant immediately upon generating aerosol. The nebulisation will continue until the chamber is empty, estimated 15 minutes, unless otherwise indicated, such as adverse event.
  The nurse/investigator will undertake clinical observations including heart rate, respiratory rate, SpO2 and blood pressure, every 5 minutes during nebulisation and then at 30 minutes, 1 hour and 2 hours. Cardiorespiratory auscultation will occur at the end of nebulisation and prior to discharge.
  This will be repeated once daily for three consecutive days.
  Blood tests will be taken before the first dose is given on day 1, and two hours after the last dose is given on day 3.
  Interventions: Drug: BromAc
- Bromac (150ug/20mg) (Experimental): The nurse/investigator will fill the jet nebuliser canister supplied on the ward with the 5ml of BromAc (150micrograms bromelain and 20mg acetylcysteine). The cannister will be collected to the mask and attached to the wall compressed air supply, with flow of between 6-8L per minute. The mask will be placed on the participant immediately upon generating aerosol. The nebulisation will continue until the chamber is empty, estimated 15 minutes, unless otherwise indicated, such as adverse event.
  The nurse/investigator will undertake clinical observations including heart rate, respiratory rate, SpO2 and blood pressure, every 5 minutes during nebulisation and then at 30 minutes, 1 hour and 2 hours. Cardiorespiratory auscultation will occur at the end of nebulisation and prior to discharge.
  This will be repeated once daily for three consecutive days.
  Blood tests will be taken before the first dose is given on day 1, and two hours after the last dose is given on day 3.
  Interventions: Drug: BromAc
- Bromac (200ug/20mg) (Experimental): The nurse/investigator will fill the jet nebuliser canister supplied on the ward with the 5ml of BromAc (200 micrograms bromelain and 20mg acetylcysteine). The cannister will be collected to the mask and attached to the wall compressed air supply, with flow of between 6-8L per minute. The mask will be placed on the participant immediately upon generating aerosol. The nebulisation will continue until the chamber is empty, estimated 15 minutes, unless otherwise indicated, such as adverse event.
  The nurse/investigator will undertake clinical observations including heart rate, respiratory rate, SpO2 and blood pressure, every 5 minutes during nebulisation and then at 30 minutes, 1 hour and 2 hours. Cardiorespiratory auscultation will occur at the end of nebulisation and prior to discharge.
  This will be repeated once daily for three consecutive days.
  Blood tests will be taken before the first dose is given on day 1, and two hours after the last dose is given on day 3.
  Interventions: Drug: BromAc

INTERVENTIONS:
Drug: BromAc — Bromelain and acetylcysteine are combined in various concentrations (either 100ug, 150ug or 200ug of bromelain, with 20mg of acetylcysteine). This is then delivered by a nebuliser to up to 12 healthy volunteers. The primary aim is determining safety.

SUMMARY:
COVID-19 is a disease that has multiple facets including an inflammatory storm, it promotes blood clotting and causes kidney damage, mucinous secretions in the lung are of great importance to outcome. Increasingly sticky sputum is associated with critical illness, with considerably raised levels of a specific type of mucous protein (MUC5AC) in sputum in COVID-19 patients. There is a strong link between viral infection and mucus production via multiple inter-cellular signalling pathways including Interleukin (IL)6, IL10 and Tumour Necrosis Factor (TNF) whereby the inflammatory storm causes sudden secretion of high volumes of dense mucus.

An Australian pharmaceutical company has developed BromAc (Bromelain & Acetylcysteine) for the palliative treatment of highly mucinous tumors of the appendix and lung. During pre-clinical development, they found that BromAc® rapidly dissolved and removed tumour mucin, making it a potent mucolytic. In combination, bromelain and acetylcysteine disrupt the architecture of the SARS-COV-2 virus in a way that renders it non-infective, reduced cytokines and chemokines in COVID-19 sputum and is a highly effective respiratory mucolytic.

The aim of this study is to assess whether BromAc delivered into the respiratory tract as a nebulised aerosol is tolerated and safe at three specific concentrations in healthy volunteer participants. The investigators will further assess the safety of nebulised BromAc and efficacy of the drug product as a mucolytic and anti-inflammatory, and whether this improves clinical outcome in participants with COVID-19. The hypothesis is that BromAc will be tolerated by patients and will result in mucus clearance, improving oxygenation and compliance in those that are ventilated.

This is a phase I study on the safety of BromAc, where 12 healthy volunteers will receive BromAc as a nebulised aerosol into the respiratory tract. BromAc is a product that combines two existing products to be delivered into the respiratory tract via nebulised aerosol delivery through a mask. The participant will be assessed for symptoms and side effects. The participant will receive nebulised BromAc at the allocated dose level for a total of 3 days. The hypothesis is that nebulised airway delivery of BromAc will be safe at the concentrations assessed.

DETAILED DESCRIPTION:
The SARS-CoV-2 virus, with its clinical syndrome known as COVID-19, has a spike protein (S), nucleocapsid protein (N) that contains the RNA, membrane protein (M) and the envelope protein (E). The spike protein is responsible for initiating internalisation of the virus genome into human lung cells via ACE2 receptors in the nasopharyngeal and lung tissue, it protrudes on the outer surface and is made up of number of amino acids and glycoproteins. The integrity of the proteins (S, N, M & E) is vital for viral functions, and formation of disulfide bonds between these have been suggested to play a vital role in the performance of the protein. The cleavage site after binding has been reported to split the spike glycoprotein, which is then reported to be supported with disulphide bonds. Binding then triggers proteolysis processed by transmembrane protease, serine 2 (TMPRSS2), furin, and perhaps other proteases, leading to fusion of viral and cellular membranes and thus target cells penetration. Hijacking of the cellular machinery then allows viral multiplication.

COVID-19 is a disease that has multiple facets including cytokine storm, thromboembolism and renal impairment, but the investigators believe mucinous secretions in the lung are of great importance to outcome. Early reports of lung pathology included cellular fibromyxoid exudate, proteinaceous exudate, massive luminal fibrous exudate and severe mucoid tracheal bronchitis. Autopsies in a cohort of fatal cases from northern Italy showed 'lumina often contained dense mucoid material. There are many pathological changes in the lungs, and these evolve over time. Early disease is characterised by neutrophilic exudative capillaritis with thrombosis. Late changes occurring on average from day 10 include diffuse alveolar damage, intravascular thrombosis, infection, disseminated intravascular coagulopathy (DIC) and later intra-alveolar fibroblast proliferation. Bronchoscopy was performed for acute hypoxia due to lung collapse in a COVID-19 patient, revealing a thick mucus plug. Multiple other reports of similar findings in bronchoscopies have been described where mucolytic therapy and suctioning have been advocated. Sputum characteristics in patients with severe COVID-19 correlate with outcome. Increasingly sticky sputum was associated with critical illness and considerably raised levels of MUC5AC in sputum in COVID-19 patients. There is a strong link between viral infection and mucus production via multiple signalling pathways including Interleukin (IL)6, IL10 and Tumour Necrosis Factor (TNF) whereby the cytokine storm causes sudden mucus hypersecretion.

Currently, there are few therapeutic agents of limited efficacy to treat or avoid the complications of COVID-19. An Australian pharmaceutical company has developed BromAc for the palliative treatment of highly mucinous tumors of the appendix and lung. This drug is composed of bromelain and acetylcysteine. During pre-clinical development, the sponsor found that BromAc® rapidly dissolved and removed tumour mucin, making it a potent mucolytic. BromAc® in combination have the ability, as shown in pre-clinical studies, to remove the mucin protective framework expressed by cancer including mucins MUC1, MUC2, MUC4, MUC5AC and MUC16. The sponsor has that BromAc breaks peptide and glycosidic linkages and disulphide bonds in tumour produced and respiratory mucin. It also combines synergistically with a variety of anticancer and antibacterial drugs.

In an in vitro study with Vero and CALU-3 cells infected by SARS-CoV-2 (MOI 1 to -4) and treated with BromAc, it was found that the drug was able to reduce the virus' ability to infect cells, demonstrating an antiviral potential against SARS-CoV-2. In addition to the anti-viral effect, BromAc is a potent mucolytic. In laboratory studies conducted in Brazil, BromAc (125ug or 250ug/ml plus 20mg/ml Acetylcysteine) resulted in complete dissolution of severe COVID-19 sputum within 30 minutes. BromAc was also shown to significantly down-regulate cytokines and chemokines in comparison to Acetylcysteine alone or control, specifically those important to COVID-19 cytokine storm CCL2, CCL3, IL-6, CXCL10. In vitro safety models have received nebulised and intranasal BromAc up to 500ug/20mg/ml three times daily for five days, with no evidence of toxicity.

In oncology, BromAc interferes with the effect of mucin, reduces cancer cell viability and profoundly enhances the effects of certain chemotherapy agents. MUC1, MUC2 and MUC5AC are highly expressed in gastrointestinal tumours. In brief, when investigating the effects of BromAc treatment on specific mucin isoforms in gastrointestinal carcinoma cells, the sponsor observed a significant decrease in the expression of MUC2 and MUC5AC in gastrointestinal LS174T cell lines. MUC1 and MUC5 are overexpressed and aberrantly glycosylated in most carcinomas, exploited by malignant cells to induce transformation and tumorigenicity. The sponsor's team have performed dose escalation animal safety studies with repeat injection in three different animal species into the peritoneum with doses of Bromelain up to 10mg/kg and Acetylcysteine 500mg/kg. There was no toxicity seen. BromAc was shown to remove mucin from the a range of human tumours in vivo, while none of the drugs worked alone. BromAc has the ability, as demonstrated in preclinical studies, to remove the protective structure of mucin expressed by cancer, including MUC1, MUC2, MUC4, MUC5B, MUC5AC and MUC16. BromAc's mechanism of action in removing peptide and glycoside bonds and disulfide bonds in mucin has also been shown. In addition, secondary infection in patients with COVID-19 might also be prevented or treated because of the effect of BromAc on biofilm. The sponsor has described efficacy in used endotracheal tubes at dissolving biofilm via nebulisation of BromAc, in addition to extensive laboratory work on pseudomonas aeruginosa and staphylococcus aureus established biofilms.

It is known that oxygen exchange is the main problem in patients with COVID-19 and hypoxia is one of the most serious effects, in which patients succumb to acute respiratory distress syndrome (ARDS). The development of mucinous sputum plugs in individuals infected with SARS-CoV-2 is variable in the early stages of the disease. In addition, 30-40% of patients who are in hospital have expectoration production, and in a recent study on pulmonary pathology in patients with COVID-19, subsequent tests revealed markedly increased levels of MUC1 and MUC5AC in sputum and trachea aspirate.

This study aims to examine the safety and efficacy of nebulised BromAc in a dose escalation phase I component. A phase I study applying the safe and effective dose in patients with moderate to severe COVID-19 will also be conducted. The primary endpoint in the phase I studies is the safety and tolerability of the planned doses. The hypothesis is that BromAc will be tolerated by patients and will result in mucus clearance, improving oxygenation and compliance in those that are ventilated.

This is a phase I study on the safety of BromAc, where 12 healthy volunteers who are otherwise well and remain in the outpatient setting will receive BromAc as a nebulised aerosol into the respiratory tract. BromAc is a product that combines two existing products (Bromelain and Acetylcysteine), along with 0.9% normal saline to be delivered into the respiratory tract via nebulised aerosol delivery through a mask. The participant will be assessed for symptoms and side effects.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to 70 years
* Received complete vaccination against COVID-19 over one week from trial commencement, able to adhere to Health guidelines surrounding attendance to a public hospital, and completion of any hospital questionnaires
* Are considered suitable for the trial based on ability to follow protocol and provide informed consent
* Are within a 10km radius of a study centre for ensuring adherence to trial procedures and follow up

Exclusion Criteria:

* Have been in contact with a known case of COVID-19 or advised to undertake self-isolation
* Have known allergy (anaphylaxis) or sensitivity to pineapples, papain, bromeliads, (fruit or plant) sulphur, eggs or Acetylcysteine that cannot be managed with steroids or antihistamine prophylaxis or any other serious unrelated allergy
* Have symptoms of COVID-19 such as cough or shortness of breath or evidence of pulmonary disease, other respiratory disease including asthma or chronic obstructive pulmonary disease
* Have a coagulation disorder of any kind or are on anticoagulant or anti-platelet therapy, history of nose bleeds or easy bruising
* ECOG >2
* Have any other serious comorbidities where inclusion in the trial will subject the patient to a higher risk of adverse events
* Pregnant women are excluded from this study because BromAc has unknown but a potential risk for adverse events in nursing infants secondary to treatment of the mother. Breastfeeding should be discontinued if the mother is treated with BromAc
* Patients with psychiatric illness/social situations that would limit compliance with study requirements
* Are unable to give fully informed and educated consent or are unable to comply with the standard follow up procedures of a clinical trial

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2022-07-27 (Actual); Primary Completion 2022-08-14 (Actual); Study Completion 2022-08-25 (Actual)

PRIMARY OUTCOMES:
To characterise and evaluate the safety of BromAc following nebulised delivery | Heart rate will be measured every 10 minutes during nebulisation, then 30 minutes after cessation of treatment and again at 1 hour and 2 hours.
  Clinical observations will be performed to to assess change compared to baseline in heart rate (HR) (beats per minute).
To characterise and evaluate the safety of BromAc following nebulised delivery | Blood pressure will be measured every 10 minutes during nebulisation, then 30 minutes after cessation of treatment and again at 1 hour and 2 hours.
  Clinical observations will be performed to assess change compared to baseline in blood pressure (BP) (mmHg)
To characterise and evaluate the safety of BromAc following nebulised delivery on oxygen saturation | SpO2 will be measured every 10 minutes during nebulisation, then 30 minutes after cessation of treatment, and again at 1 hour and 2 hours.
  Clinical observations will be performed to assess change compared to baseline in SpO2 (oxygen saturation) to determine SpO2 to FiO2 (fraction of inspired oxygen) ratio.
To characterise and evaluate the safety of BromAc following nebulised delivery on respiratory rate | Respiratory rate will be measured every 10 minutes during nebulisation, then 30 minutes after cessation of treatment, and again at 1 hour and 2 hours.
  Clinical observations will be performed to assess change compared to baseline in respiratory rate (RR) (breaths per minute)
To characterise and evaluate the safety of BromAc following nebulised delivery on mucosal parameters | Baseline each treatment day and at the end of each nebulisation on days 1-3.
  Mucosal assessment will be performed by the Total Nasal Symptom Score to determine any changes in mucosal parameters vs baseline. A higher score will mean a worse outcome in terms of nasal mucosal side effect to treatment.
To characterise and evaluate the safety of BromAc following nebulised delivery on blood parameters | Blood tests will be performed at baseline (day 0), then each day of treatment (days 1-5), during follow up on day 6 and day 14.
  Biochemical analyses liver and kidney function, full blood count, coagulation and inflammatory markers will be measured and compared to baseline pretreatment results to determine if there is any change to the baseline biochemical parameters of the drug treatment.

SECONDARY OUTCOMES:
Determine the proportion of patients with treatment-emergent adverse events (AEs) | Adverse events will be monitored during and immediately post-treatment on days 1, 2 and 3; and for delayed adverse events on days 4, 5 and 10 and 14.
  Any adverse drug effects (ADE) using the FDA safety guidance for healthy volunteer criteria including nausea/vomiting, diarrhoea, fatigue, myalgia, headache, or any other bodily discomfort.
Determine the maximum tolerated dose (MTD) of BromAc within he therapeutic range for COVID-19 delivered by nebuliser | At each dose escalation and up until the end of follow up (last day of follow up for the last patient enrolled).
  At each dose level (100ug, 150ug and 200ug bromelain), safety/toxicity will be monitored and progression onto the next level will be decided pending an appropriate safety profile

CONTACTS AND LOCATIONS:
Overall Officials: Frank van Haren, MD, PhD, Principal Investigator — St George Hospital, Director of Intensive Care
Locations (1):
- St George Hospital, Kogarah, New South Wales, Australia